CLINICAL TRIAL: NCT03868137
Title: Multi-dose Ibuprofen Prophylaxis for IUD-insertion (MIPI): A Triple Blinded
Brief Title: Multi-dose Ibuprofen Prophylaxis for IUD-insertion
Acronym: MIPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orlando VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chensi Ouyang, Physician, Orlando VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1335793-1
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Pelvic Pain; IUD
Keywords: NSAID; Intrauterine Devices; Ibuprofen; Pelvic pain
MeSH Terms: conditions — Pelvic Pain | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Triple blind randomized control trial involving placebo arm and intervention arm (Ibuprofen)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization sequence will be generated and given to the research pharmacist who will dispense the appropriate medications to the participants in each arm. Only the pharmacist will know which patient is in which trial arm until the study has ended and data has been analyzed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 3 doses of placebo identical to study drug will be given to patients starting 1 day before IUD insertion
  Interventions: Drug: Placebos
- Ibuprofen (Experimental): 3 doses of Ibuprofen 800 mg will be given to patients starting 1 day before IUD insertion. Patient will take 800 mg Ibuprofen at noon and 8 PM day before IUD insertion and at 8 AM on the day of IUD insertion.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — 3 doses of Ibuprofen 800 mg
  Arms: Ibuprofen
Drug: Placebos — Placebo
  Arms: Placebo

SUMMARY:
This study compares the effectiveness of decreasing pain at time of and day after intrauterine device (IUD) insertion when patients take three doses of Ibuprofen versus three doses of placebo.

DETAILED DESCRIPTION:
Ibuprofen is commonly used over the counter and prescribed for pain relief such as menstrual cramps. Intrauterine (IUD) insertion can cause pain during and after the insertion. Currently, studies have found that single dose of Ibuprofen take prior to IUD insertion does decrease pain at time of IUD insertion. This study will examine whether 3 doses of Ibuprofen can decrease pain at time of and 1 day after IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Female
* Able to provide informed consent
* English speaking
* Able to provide telephone and address contact information
* Able and willing to receive HIPAA compliant telephone texts and phone messages
* Stable (the same) address and phone number within the last 6 months.

Exclusion Criteria:

* Contraindications to IUD insertion (active pelvic infection, current pregnancy)
* Contraindications to NSAIDs (allergy, history of asthma, history of aspirin allergy, history of kidney disease, history of stomach ulcer, history of active GI bleeding, history of liver disease)
* Not undergoing any other concurrent office procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient must be female since IUDs are female contraception.
Enrollment: 86 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Pain at time of IUD insertion | At time of IUD insertion
  Pain score measured on 10 point visual analog scale (VAS): 0-3 mild pain, 4-7 moderate pain, 8-10 severe pain

SECONDARY OUTCOMES:
Pain at 1 day after IUD insertion | 1 day after IUD insertion
  Pain score measured on 10 point visual analog scale (VAS): 0-3 mild pain, 4-7 moderate pain, 8-10 severe pain
Usage of other medications or methods to decrease post-IUD insertion pain | 1 day after IUD insertion
  Names of other medications or methods

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando VA Medical Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kavanaugh ML, Jerman J, Finer LB. Changes in Use of Long-Acting Reversible Contraceptive Methods Among U.S. Women, 2009-2012. Obstet Gynecol. 2015 Nov;126(5):917-927. doi: 10.1097/AOG.0000000000001094. PMID 26444110
- [Background] Asker C, Stokes-Lampard H, Beavan J, Wilson S. What is it about intrauterine devices that women find unacceptable? Factors that make women non-users: a qualitative study. J Fam Plann Reprod Health Care. 2006 Apr;32(2):89-94. doi: 10.1783/147118906776276170. PMID 16824298
- [Background] Hubacher D, Reyes V, Lillo S, Pierre-Louis B, Zepeda A, Chen PL, Croxatto H. Preventing copper intrauterine device removals due to side effects among first-time users: randomized trial to study the effect of prophylactic ibuprofen. Hum Reprod. 2006 Jun;21(6):1467-72. doi: 10.1093/humrep/del029. Epub 2006 Feb 16. PMID 16484309
- [Background] Jensen HH, Blaabjerg J, Lyndrup J. [Prophylactic use of prostaglandin synthesis inhibitors in connection with IUD insertion]. Ugeskr Laeger. 1998 Nov 23;160(48):6958-61. Danish. PMID 9846090
- [Background] Chor J, Bregand-White J, Golobof A, Harwood B, Cowett A. Ibuprofen prophylaxis for levonorgestrel-releasing intrauterine system insertion: a randomized controlled trial. Contraception. 2012 Jun;85(6):558-62. doi: 10.1016/j.contraception.2011.10.015. Epub 2011 Dec 15. PMID 22176793
- [Background] Bednarek PH, Creinin MD, Reeves MF, Cwiak C, Espey E, Jensen JT; Post-Aspiration IUD Randomization (PAIR) Study Trial Group. Prophylactic ibuprofen does not improve pain with IUD insertion: a randomized trial. Contraception. 2015 Mar;91(3):193-7. doi: 10.1016/j.contraception.2014.11.012. Epub 2014 Nov 25. PMID 25487172
- [Background] Massey SE, Varady JC, Henzl MR. Pain relief with naproxen following insertion of an intrauterine device. J Reprod Med. 1974 Dec;13(6):226-31. No abstract available. PMID 4612152
- [Background] Ngo LL, Ward KK, Mody SK. Ketorolac for Pain Control With Intrauterine Device Placement: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):29-36. doi: 10.1097/AOG.0000000000000912. PMID 26241253
- [Background] Ngo LL, Braaten KP, Eichen E, Fortin J, Maurer R, Goldberg AB. Naproxen Sodium for Pain Control With Intrauterine Device Insertion: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1306-1313. doi: 10.1097/AOG.0000000000001746. PMID 27824753
- [Result] Trussell J. Contraceptive failure in the United States. Contraception. 2011 May;83(5):397-404. doi: 10.1016/j.contraception.2011.01.021. Epub 2011 Mar 12. PMID 21477680
- [Result] Lethaby A, Hussain M, Rishworth JR, Rees MC. Progesterone or progestogen-releasing intrauterine systems for heavy menstrual bleeding. Cochrane Database Syst Rev. 2015 Apr 30;(4):CD002126. doi: 10.1002/14651858.CD002126.pub3. PMID 25924648